CLINICAL TRIAL: NCT04508998
Title: Mechanistic Study of the Effect of ET-1 SNPs in Coronary Microvascular Disease
Brief Title: PRIZE ET Sub-Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P02664
Record Dates: First submitted 2020-06-21; First posted 2020-08-11 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Microvascular Angina
Keywords: angina; endothelin receptor antagonist; zibotentan
MeSH Terms: conditions — Microvascular Angina; Angina Pectoris | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with microvascular angina (Experimental): Patients with clinical features of microvascular angina screened for the main PRIZE trial however not possessing the PHACTR1 GG minor allele single nucleotide polymorphism
  Interventions: Diagnostic Test: Blood tests including genotyping; Diagnostic Test: Exercise Tolerance Test

INTERVENTIONS:
Diagnostic Test: Blood tests including genotyping — Blood tests for alternative SNPs altering levels of ET-A receptor expression; blood will be further analysed for endothelin receptor mRNA and other plasma peptides important in the endothelin signalling pathway
Diagnostic Test: Exercise Tolerance Test — Treadmill exercise test using the Bruce protocol

SUMMARY:
Microvascular angina (MVA) is caused by abnormalities of the small blood vessels in the heart. Endothelin-1 (ET-1) is a chemical messenger that circulates and accumulates in the blood vessel walls, causing them to narrow or go into spasm and thicken over a long period, especially as levels of ET-1 increase. As a result, patients experience pain, psychological distress and limitation of their daily activities.

Cambridge is a participating recruitment site for a large randomised, double blinded, placebo controlled crossover trial (the PRIZE study: NCT04097314) investigating Zibotentan as a new drug treatment for patients with MVA using a 'precision medicine' approach. Zibotentan is a drug originally developed by Astra Zeneca for prostate cancer but prior research has shown that it acts to relax the small blood vessels of patients with MVA, highlighting its potential as a novel therapy for this patient group. The PRIZE study population will be enriched for 'responders' to the drug by screening patients with MVA for a gene mutation known to increase levels of circulating endothelin. The trial aims to initially invite approximately 356 participants for genetic testing but only 100 participants will go forward into the main study, with approximately 2/3rd being screen failures.

In our sub-study, we will invite patients with MVA who are screen failures at our site for further blood tests looking for other genetic variants in the ET-1 signalling pathway and examine how this correlates with the severity of microvascular angina quantified by cardiac MRI and clinical assessments. Data from this sub-study would provide a bio-resource for further analysis of the main PRIZE trial to identify other patients that would benefit from Zibotentan.

DETAILED DESCRIPTION:
Patients with microvascular angina (MVA) are under-diagnosed and have limited therapeutic options available to them. Endothelin-1 (ET-1) is a potent vasoconstrictor implicated in the small vessel obstruction that causes MVA. The PRIZE trial will apply a precision medicine approach to assess the therapeutic effect of Zibotentan, an ET-1 antagonist (ETA) selective for the ETA receptor in patients who are high ET-1 expressors (possessing the PHACTR1 minor GG allele single nucleotide polymorphism - SNP). Unfortunately, the incidence of this SNP occurs in only a third of the population, resulting in a high screen-failure rate.

In the proposed sub-study, we aim to recruit patients with MVA but without the minor GG allele SNP to potentially identify other potential 'responders' to Zibotentan. In an observational mechanistic study, we will perform baseline genotyping for other genetic variants in the ET-1 pathway as well as phenotyping patients by quantification of microvascular disease from retrospective analysis of cardiac MRI data. Patients will also complete angina and quality of life questionnaires and perform an exercise stress test to determine maximal exercise distance. Information from this sub-study will provide a genotype bio-resource that could identify novel SNPs for the pathogenesis of MVA that could be validated in the UK biobank. This may indicate other ETA receptor antagonist super-responders, justifying treatment with Zibotentan and enabling more patients with MVA to potentially benefit from this promising drug.

ELIGIBILITY:
Patients who after screening blood tests and clinical assessment are ineligible for the main PRIZE trial will qualify for this study. Patients will be screened for the PRIZE trial according to the following:

Inclusion criteria:

1. Age >18 years.
2. Probable or definite Microvascular Angina as defined in COVADIS criteria:

   * Clinical symptoms of angina
   * No obstructive coronary artery disease
   * Objective evidence of myocardial ischemia
   * Evidence of impaired coronary microvascular function (Optional)
3. Able to comply with study procedures.
4. Screen failure for the main PRIZE study
5. Written informed consent.

Exclusion criteria:

1. Lack of informed consent for the PRIZE ET Sub-study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2022-08-13 (Actual)

PRIMARY OUTCOMES:
Correlation of ET-A SNPs with ET-A expression in blood by qPCR, levels of endothelin related plasma peptides and clinical data (exercise duration and microvascular disease measured by quantitative perfusion on Cardiac MRI) | correlation will be assessed at baseline at the start of the trial (time point 0)
  Measurement of molecules associated with the endothelin signalling pathway in patients with different SNPs for the ET-A receptor will be compared with phenotypic characteristics of the patients, specifically exercise tolerance and by retrospective analysis of the patient's cardiac MRI using quantitative measures of myocardial blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hoole, Principal Investigator — Royal Papworth NHS Foundation Trust
Locations (1):
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be entered on electronic clinical record forms inputed on the Open Clinica eCRF platform with password protected access for researchers and for quality assurance personnel only.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: A combined analysis with other leftover patient samples from other PRIZE trial participating sites is in progress. It is anticipated the clinical study report will be available in February 2024
Access Criteria: Individual participant data will not be shared routinely in this or any related research.

REFERENCES:
- [Background] Abraham GR, Morrow AJ, Oliveira J, Weir-McCall JR, Davenport EE, Berry C, Davenport AP, Hoole SP. Mechanistic study of the effect of Endothelin SNPs in microvascular angina - Protocol of the PRIZE Endothelin Sub-Study. Int J Cardiol Heart Vasc. 2022 Feb 25;39:100980. doi: 10.1016/j.ijcha.2022.100980. eCollection 2022 Apr. PMID 35242999
- See also: Related Info — https://doi.org/10.1016/j.ijcha.2022.100980